CLINICAL TRIAL: NCT03529838
Title: Hemodynamic Responses and Salivary Markers of the Interaction of 12 Weeks of Training With Different Anti-hypertensive in Menopausal Women
Brief Title: Hemodynamic and Salivary Responses of 12 Weeks of Training With Different Anti-hypertensive
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Early interruption caused by the COVID-19 pandemic.
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Igor Moraes Mariano, Bachelor, Federal University of Uberlandia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 71285317.4.0000.5152
Record Dates: First submitted 2018-05-08; First posted 2018-05-18 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Hypertension; Menopause
Keywords: Combined Exercise; Ambulatorial Blood Pressure Monitoring; Blood analysis; Salivary analysis; Heart rate variability
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: 45 women taking different antihypertensives (15 no medications, 15 angiotensin receptor blockers and 15 beta blockers) for at least 6 months will be assessed at baseline and after 12 weeks of combined exercise training.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No medication (Placebo Comparator): Group of pre-hypertensive women with no medication who practiced 12 weeks of training with Combined Exercise Training, non-obese, nonsmokers and with no characteristics that prevented them from performing the activities. In addition this group could not modify the dose or type of the medicine and should be using the same medicine and dose for at least 6 months
  Interventions: Other: Combined exercise
- Angiotensin receptor blockers (Active Comparator): Group of hypertensive women taking Angiotensin receptor blockers who practiced 12 weeks of training with Combined Exercise Training, non-obese, nonsmokers and with no characteristics that prevented them from performing the activities. In addition this group could not modify the dose or type of the medicine and should be using the same medicine and dose for at least 6 months
  Interventions: Other: Combined exercise
- Beta blockers (Active Comparator): Group of hypertensive women taking Beta blockers who practiced 12 weeks of training with Combined Exercise Training, non-obese, nonsmokers and with no characteristics that prevented them from performing the activities. In addition this group could not modify the dose or type of the medicine and should be using the same medicine and dose for at least 6 months
  Interventions: Other: Combined exercise

INTERVENTIONS:
Other: Combined exercise — The program consisted of 36 sessions of combined aerobic and resistance exercises training during 12 consecutive weeks. Each session lasted 60 minutes and consisted of 30 minutes of resistance exercise and 30 minutes of aerobic exercise. The resistance training was performed in two sets of 8 to 12 repetitions in five exercises of weight training (Based on 1 repetition maximum test - 1RM). The aerobic exercise was performed on a treadmill, at a speed of 5.5 km/h and intensity (imposed by treadmill inclination and heart rate) between 65 and 75% of maximun heart rate measured in maximum incremental test. Every week the resistance load and aerobic intensity was readjusted by determined training zone (8 to 12 maximum repetitions) and heart rate predicted in the incremental respectively.

SUMMARY:
Different classes of antihypertensives may have different responses when associated with exercise. Thus, this study aims to compare the responses of the association of 12 weeks of aerobic exercise and weightlifting with different classes of medications in 45 postmenopausal hypertensive women.

DETAILED DESCRIPTION:
Cardiovascular diseases are the leading causes of death and postmenopausal women. Physical exercise, in turn, is a strategy to reduce cardiovascular stress, by decreasing the blood pressure (BP) at rest and several risk factors associated with sedentary lifestyle, thus improving the quality and life expectancy of these women. However, different classes of antihypertensives may have different responses when associated with exercise. Thus, this study aims to compare the responses of the association of 12 weeks of aerobic exercise and weightlifting with different classes of medications in 45 postmenopausal hypertensive women. The volunteers will do cardiovascular and biochemistry evaluations before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 50 and 70 years;
* Be in the postmenopausal phase;
* Be able to practice physical exercise on treadmill and bodybuilding,
* Receive a release certificate for exercise practice;
* Do not present physical problems or cardiovascular complications that prevent the performance of physical exercises;
* In the case of hypertensives: present stage 1 hypertension, according to the guidelines of the Brazilian Society of Hypertension (2010);
* In the case of hypertensive patients, undergo drug treatment with β-blockers or Angiotensin receptor blockers.

Exclusion Criteria:

* Present history of stroke or acute myocardial infarction;
* Smokers;
* Present diagnosis of Diabetes Mellitus or renal pathologies;
* Use of antihypertensive drugs from classes that were not selected for this project;
* Make use of hormonal therapies;
* Being uncompensated hypertensive.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Changes in Ambulatorial Blood Pressure | Before and within 72 hours after 12 weeks of exercise training
  All volunteers were submitted to a 24-hour Blood Pressure (BP; systolic and diastolic measurements) assessment by Ambulatorial Blood Pressure Monitoring (ABPM) before and after 10 weeks of combined exercise training, with a minimum of 48 hours after the last training session. A device was used associated with a diary of examination to self-report of activities of daily living (sleep, work, food) or any event that could interfere abnormally with BP or device measurements. The device was always placed 7am and the measurements were made every 15 minutes from 7h to 23h and every 30 minutes from 23h to 7h. The monitoring was considered valid when it happened for a period of 24 hours. The following results were evaluated: systolic blood pressure; diastolic blood pressure, mean blood pressure and heart rate in awake, sleep and 24-hour periods. Before the use ABPM during daily activities, resting blood pressure were measured using the same equipment after 15 min of rest in siting position.

SECONDARY OUTCOMES:
Changes in Ambulatorial Blood Pressure Variability | Before and within 72 hours after 12 weeks of exercise training
  Based on Ambulatorial Blood Pressure data, were calculated Blood Pressure Variability by: 24-hour standard deviation weighted by the time interval between consecutive readings; the mean diurnal and nocturnal deviations weighted for the duration of the daytime and nighttime interval; the average real variability weighted for the time interval between consecutive readings; the ambulatory arterial stiffness index calculated by the slope of the trend curve of the dispersion of pressure data; the morning surge that represents the dynamic daytime variation in morning pressure that tends to increase, being assessed from the point of least pressure during sleep in relation to the first two hours after waking; and nocturnal dipping, that represents the average percentage drop of sleep pressure in relation to wakefulness, and individuals with falls of 10% or more are considered dippers and below that are considered nom-dippers.
Changes in Heart Rate Variability | Before and within 72 hours after 12 weeks of exercise training
  Heart Rate (HR) was recorded using a heart rate monitor in a beat-by-beat basis. HR was registered in a seat position for 20 min of rest. Prior to the HR Variability (HRV) analysis, the RR intervals (RRi) were visually inspected and filtered using a moving average filter. The HRV was analyzed in both time-, frequency- and nonlinear-domain. Being that for frequency-domain analysis, firstly the RRi series were interpolated at 4 Hz and then the signal linear trend component removal was performed using the smooth priors approach.
Changes in salivary oxidative stress | Before and within 72 hours after 12 weeks of exercise training
  The salivary was collected after 12-hours fasting and the total antioxidant capacity was evaluated using the Ferric-Ability of Plasma (FRAP) methodology and calculated from the standard trolox curve. The activity of the enzyme superoxide dismutase (SOD) was determined based on the auto oxidation capacity of pyrogallol and catalase activity (CAT) by monitoring the consumption of hydrogen peroxide at 240 nm. Lipid peroxidation levels were determined by the TBARS method (thiobarbituric acid reactive substances), using as standard a curve of 1,1,3,3-tetraethoxypropane (TMP). The total protein concentration was obtained using bovine serum albumin (BSA) as standard. The amounts of nitric oxide (NO) were estimated by the determination of total nitrite by the Griess colorimetric method.
Changes of blood pressure reactivity | Before and within 72 hours after 12 weeks of exercise training
  To evaluate reactivity of blood pressure under mental stress, the Stroop protocol will be used. The test consists of a video on a computer screen facing the volunteer that changes the image every 2 seconds. Then the volunteers should speak as quickly as possible the color of the letters present on the screen, and in each image there is dissonance between the background color, the color of the letters and the word formed (which is always the name of another color). Each minute of the test the blood pressure (systolic and diastolic) will be measured by auscultatory method. To evaluate the reactivity of blood pressure under physical stress will be used the Cold pressor test. The test consists of immersing the volunteers' right hand for 1 minute in water maintained at 4ºC. Blood pressure is then assessed in the left arm after 30 and 60 seconds of immersion and after 2 minutes after the end of immersion in water. The blood pressure measurements will be done by auscultatory method.
Changes of Biochemical markers on blood | Before and within 72 hours after 12 weeks of exercise training
  Venous blood samples will be collected with 12 hours of fasting. After local asepsis, 10 ml of blood will be obtained at each collection through the puncture of the ulnar or radial ulnar vein, using a syringe and disposable needles. The blood samples will be deposited in test tubes containing ethylenediamine tetraacetic acid (EDTA) and dried tubes with separator gel for collection of serum. The samples will then be centrifuged at 2000 rpm for 15 minutes to separate plasma and serum aliquots and stored at -80 ° C for further biochemical analysis. Thus, the samples will be analyzed in the following variables: Lipid Profile, Superoxide Dismutase (SOD), Catalase (CAT), Thiobarbituric Acid (TBARS), Nitrite/nitrate (NOx-), Interleukin-6 (IL-6), Interleukin-10 IL-10), Interleukin-1 beta (IL-1b), Tumor Necrosis Factor alpha (TNFa), Creatine Kinase (CK), C-reactive protein (P-CR) and Adiponectin.

CONTACTS AND LOCATIONS:
Locations (1):
- Guilherme Morais Puga, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mariano IM, Amaral AL, V Carrijo VH, Costa JG, Rodrigues ML, Cunha TM, Puga GM. Different cardiovascular responses to exercise training in hypertensive women receiving beta-blockers or angiotensin receptor blockers: A pilot study. Clin Exp Hypertens. 2022 Jul 4;44(5):442-450. doi: 10.1080/10641963.2022.2065290. Epub 2022 Apr 23. PMID 35465803